CLINICAL TRIAL: NCT03622814
Title: Mealtime Partnerships for People With Dementia in Respite Centers and at Home
Brief Title: Partners at Meals - Respite Care and Home (PAM)
Acronym: PAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00064441
Record Dates: First submitted 2018-05-03; First posted 2018-08-09 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Dementia, Alzheimer Type; Weight Loss
Keywords: caregiving; mealtimes; respite care; train-the-trainer
MeSH Terms: conditions — Alzheimer Disease; Weight Loss

STUDY DESIGN:
Intervention Model Description: A randomized cluster-design trial will be conducted in two large respite care centers (RCCs) with five sites that serve primarily white and African American persons with dementia. RCCs were randomized to the intervention condition (Partners at Meals; 3 sites) or ['enhanced usual care' (EUC)] (2 sites). The primary unit of analysis is the person with dementia (PWD) and caregiver (CG).
Who Masked: Participant
Masking Description: Participants did not know if they are in a site that is receiving the treatment or in the usual condition site. Randomization is by site, not by individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment - Partners at Meals (PAM) (Experimental): People with dementia (PWD) often lose weight and suffer subsequent health issues: the goal of this intervention was to improve or maintain weight of a PWD, and to improve or maintain food intake. A train-the-trainer intervention is used with volunteers in Respite Care Centers who partner with family caregivers of PWD. Designed to be personalized to the PWD and focusing on his/her existing strengths and compensating for his/her deficits in mealtime management, sessions occur initially (1 hr) and every month (~30 mins) to reinforce key areas of behavioral or environmental change. Samsung tablets were used initially and then monthly (x5) to record mealtimes in the home, and were reviewed by the volunteer with the family member at the monthly session to discuss areas where changes could be made. Weight of the PWD was measured initially and monthly (x5).
  Interventions: Behavioral: Partners at Meals
- Enhanced Usual Condition (EUC) (Placebo Comparator): In the non-treatment respite care centers, an Enhanced Usual Condition was delivered to caregivers of People with Dementia (PWD). This program consisted of enhanced training in caregiving using components from a module of the evidence-based Savvy Caregiver program (K. Hepburn) given in a group setting with opportunity for a question and answer period; the program is given for new enrollees and every 6 months. The PI (TK), the nutritionist (KM) or the Program Manager (MCP) lead these groups. Weight of the PWD was measured initially and monthly (x5).
  Interventions: Behavioral: Enhanced Usual Condition

INTERVENTIONS:
Behavioral: Partners at Meals — The focus of the intervention was to facilitate meals using knowledge of the person with dementia's past history and lifelong preferences as well as their stage of disease, altering the behavior of the caregiver at meals to ameliorate dysfunctional behaviors, and altering the environment to make it more focused on the process of meals. Families recorded three meals including behavior at home each month.
  Other Names: PAM
  Arms: Treatment - Partners at Meals (PAM)
Behavioral: Enhanced Usual Condition — Enhanced Usual Condition (EUC) Staff and volunteers at the EUC sites received training in communication between family and friends of the person with dementia. Following the general model of the Savvy Caregiver (Hepburn), communication training will occur every six months in these two sites. Families will be trained by project staff to record three meals including behavior at home each month.
  Other Names: EUC
  Arms: Enhanced Usual Condition (EUC)

SUMMARY:
The goal of this study was to test the efficacy of a mealtime intervention in respite care centers for people with dementia and their caregivers. Mealtimes become more challenging as dementia progresses causing nutritional and behavioral issues in the affected individuals. Using a train-the-trainer program built on the Partners at Meals model, volunteers in respite centers partner worked with caregivers and developed a mealtime plan that builds on the strengths of the person with dementia (PWD), and developed a supportive environment for change. A tele-health component was involved in the communication between the respite center volunteers/staff and families. Recruitment was limited to people attending the particular respite centers. Two large RCCs with a total of 5 sites of care in suburban and rural areas of SC were the sites of this project.

DETAILED DESCRIPTION:
The goal of this study was to test the efficacy of a mealtime intervention (Partners at Meals) in respite care centers (RCCs) that provided a social model of care for people with dementia living in the community and support for their caregivers. Largely staffed by long-time volunteers, these centers support caregivers' ability to maintain their loved one in the home. Traditionally, support for social activities and mealtime offered by the RCCs cannot be extended to home. In this project, we used a telehealth interface to provide consultation to family caregivers in the context of home where problems arise.

The primary unit of analysis was PWD and their caregiver (CG) outcomes which included: a) PWD weight; b) dysfunctional behaviors at meals; c) quality of life (QOL) of both persons with dementia and their caregivers; and, d) CG self efficacy of managing meals at home.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Dementia (PWD): aged ≥ 60 years; attending a participating respite care center (RCC) at least once/week; living with or within the same property as caregiver (CG); diagnosis of Alzheimer's disease or related dementia with mild to moderate stage as demonstrated by the Functional Assessment Staging Scale (FAST) of 5 or greater and a MMSE of 12 or above; absence of wasting disorders (e.g., HIV/AIDS, heart or renal failure or COPD, end-stage cancer); some supervision required or dysfunctional behavior present (e.g., redirection)
* Caregiver (CG): lives with or on same property as the PWD; provides 4 hours or more of care/day; assists with ADLs including meals
* Volunteer: present at the RCC at least weekly (at least 4 hours/week); identify as comfortable in the teacher/coach role, and demonstrate ability to use televideo and photograph.

Exclusion Criteria:

* Persons with Dementia (PWD): not receiving enteral feeding or active treatment by a speech pathologist/therapist; not diagnosed with dysphagia as identified by caregiver or on RCC Intake Sheet. Those enrolled in or qualifying for hospice will not be included.
* Caregiver (CG): paid for services as caregiver; unable to speak or read English
* Volunteer: unable to read and speak English

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Kelechi, Principal Investigator — MUSC College of Nursing
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other investigators who have IRB approved studies; data will be anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be shared as approved by the MUSC IRB and from one year after the study closes to five years after the study closes or as long as the Principle Investigator(s) are employed by the University.
Access Criteria: Contact the PIs through the College of Nursing

REFERENCES:
- [Background] Amella Krug EJ, Qanungo S, Martin KL, Mueller M, Madisetti M, Kelechi TJ. A cluster randomized controlled trial to assess the efficacy of a telehealth-based train-the-trainer mealtime intervention delivered by respite care center volunteers to caregivers of persons with dementia to improve nutritional outcomes and quality of life. BMC Nutr. 2020 Jun 24;6:24. doi: 10.1186/s40795-020-00350-x. eCollection 2020. PMID 32587748

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Using a cluster randomized controlled experimental design based on each Respite Care Center's (RCCs; N=6) respective average monthly client census, RCCs were randomized to either the Partners at Mealtime (PAM) intervention (N=3; RCCs) or the control enhanced usual care (EUC) group (N=3; RCCs). Enrolled PWD/CG dyads were then allocated to the PAM intervention or the enhanced usual care (EUC) control groups based upon their RCC of attendance.
Units Other Than Participants: clinical sites
Groups:
- Treatment - Partners at Meals (PAM): People with dementia (PWD) often lose weight and suffer subsequent health issues: the goal of this intervention is to improve or maintain weight of a PWD, and to improve or maintain food intake. A train-the-trainer intervention is used with volunteers in Respite Care Centers who partner with family caregivers of PWD. Designed to be personalized to the PWD and focusing on his/her existing strengths and compensating for his/her deficits in mealtime management, sessions occur initially (1 hr) and every month (~30 mins) to reinforce key areas of behavioral or environmental change. Samsung tablets are used initially and then monthly (x5) to record mealtimes in the home, and are reviewed by the volunteer with the family member at the monthly session to discuss areas where changes could be made.
  Partners at Meals: The focus of the intervention is to facilitate meals using knowledge of the person with dementia's past history and lifelong preferences as well as their stage of disease, altering the behavior of the caregiver at meals to ameliorate dysfunctional behaviors, and altering the environment to make it more focused on the process of meals.
- Enhanced Usual Condition (EUC): In the non-treatment respite care centers, an Enhanced Usual Condition will be delivered to caregivers of People with Dementia (PWD). This program consists of enhanced training in caregiving using components from a module of the evidence-based Savvy Caregiver program (K. Hepburn) given in a group setting with opportunity for a question and answer period; the program is given for new enrollees and every 6 months. The PI (TK), the nutritionist (KM) or the Program Manager (MCP) will lead these groups. Weight of the PWD is measured initially and monthly (x5); amount of food consumed will be measured using the Samsung tablets, also initially and monthly (x5).
  Enhanced Usual Condition: Enhanced Usual Condition (EUC) Staff and volunteers at the EUC sites will receive training in communication between family and friends of the person with dementia. Following the general model of the Savvy Caregiver (Hepburn), communication training will occur every six months in these two sites. Families will be trained by project staff to record three meals including behavior at home each month. The Project Manager will attend the monthly support group for family members about communication. The administrator of the EUC RCC will be interviewed every 6 months the project is in place.
Period: Overall Study
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
Started | 54; 3 clinical sites | 52; 3 clinical sites
PWD | 27; 3 clinical sites | 21; 3 clinical sites
Caregiver | 27; 3 clinical sites | 21; 3 clinical sites
Completed | 46; 3 clinical sites | 38; 3 clinical sites
Not Completed | 8; 0 clinical sites | 14; 0 clinical sites
Not completed — Lost to Follow-up | 8 | 14

BASELINE CHARACTERISTICS:
Population: Participant enrollment includes caregivers and persons with dementia. While we had volunteers, they assisted with intervention delivery but we did not collect baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC) | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Categorical [Count of Participants; unit: Participants] — Population: The overall number of baseline participants includes both caregivers and persons with dementia combined.
  Participants
    Persons with dementia: number analyzed (Participants) | 27 | 26 | 53
    Persons with dementia: <=18 years | 0 | 0 | 0
    Persons with dementia: Between 18 and 65 years | 1 | 5 | 6
    Persons with dementia: >=65 years | 26 | 21 | 47
    Caregivers: number analyzed (Participants) | 27 | 26 | 53
    Caregivers: <=18 years | 0 | 0 | 0
    Caregivers: Between 18 and 65 years | 7 | 14 | 21
    Caregivers: >=65 years | 20 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data was collected from dyads which included persons with dementia (PWD) and their caregivers for both treatment and usual care arms
  years
    Persons with dementia: number analyzed (Participants) | 27 | 21 | 48
    Persons with dementia | 81.0 (7.7) | 73.9 (10.7) | 77.9 (9.2)
    Caregivers: number analyzed (Participants) | 27 | 21 | 48
    Caregivers | 69.4 (10.8) | 63.4 (12.2) | 66.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall number of baseline participants includes both caregivers and persons with dementia combined.
  Participants
    Persons with dementia: number analyzed (Participants) | 27 | 26 | 53
    Persons with dementia: Female | 13 | 10 | 23
    Persons with dementia: Male | 14 | 16 | 30
    Caregivers: number analyzed (Participants) | 27 | 26 | 53
    Caregivers: Female | 19 | 22 | 41
    Caregivers: Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number of baseline participants includes both caregivers and persons with dementia combined.
  Participants
    Persons with dementia: number analyzed (Participants) | 27 | 26 | 53
    Persons with dementia: Hispanic or Latino | 0 | 0 | 0
    Persons with dementia: Not Hispanic or Latino | 27 | 26 | 53
    Persons with dementia: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 27 | 26 | 53
    Caregivers: Hispanic or Latino | 0 | 0 | 0
    Caregivers: Not Hispanic or Latino | 27 | 26 | 53
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number of baseline participants includes both caregivers and persons with dementia combined.
  Participants
    Persons with dementia: number analyzed (Participants) | 27 | 26 | 53
    Persons with dementia: American Indian or Alaska Native | 0 | 0 | 0
    Persons with dementia: Asian | 0 | 0 | 0
    Persons with dementia: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Persons with dementia: Black or African American | 5 | 2 | 7
    Persons with dementia: White | 22 | 24 | 46
    Persons with dementia: More than one race | 0 | 0 | 0
    Persons with dementia: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 27 | 26 | 53
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 1 | 0 | 1
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 5 | 2 | 7
    Caregivers: White | 21 | 24 | 45
    Caregivers: More than one race | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Monthly Weight in Pounds on a Scale for Person With Dementia
Description: Assessed by unit of measure in pounds; reported as mean difference in pounds from baseline to follow-up at 6 months
Time Frame: This was a 6-month study. We are reporting the change from baseline to the 6-month end of study time period.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
Number analyzed (Participants) | 27 | 26
pounds | -2.1 (8.1) | -2.1 (9.9)

2. Primary Outcome: Person With Dementia: Dysfunctional Behavior at Meals Measured With the Edinburgh Feeding in Dementia Scale (EdFED)
Description: The Edinburgh Feeding in Dementia Scale (EdFED) is an observational instrument used across settings to evaluate feeding problem behavior. Using Guttmann Scaling, the EdFED Q has 4 items that measure level of assistance and 6 behavioral descriptors of specific mealtime behaviors; all are each rated 'never, sometimes, often' and cannot be rated 0, 1, 2, respectively, producing a range of 0-20 with higher scores indicating more problem behaviors. The instrument was used to also assess specific behaviors seen in moderate stage dementia such as wandering, distracted, perseverating, unable to use utensils, premature oral closure.
Time Frame: This was a 6-month study. We are reporting the change from baseline to the 6-month end of study time period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
Number analyzed (Participants) | 25 | 21
score on a scale | 4.0 (3.7) | 2.4 (6.4)

3. Primary Outcome: Person With Dementia: Quality of Life
Description: The QOL scale in Alzheimer's disease (QOL--AD) is a 13--item rating of domains of physical condition, mood, memory, functional abilities, interpersonal relationships, ability to participate in meaningful activities, financial situation, and global assessments of self as a whole and QOL as a whole. Scoring instructions for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4. The total score is the sum of all 13 items (scoring ranging from 13 to 52. Higher scores indicated better quality of life.
Time Frame: This was a 6-month study. We are reporting the change from baseline to the 6-month end of study time period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
Number analyzed (Participants) | 26 | 23
score on a scale | 33.7 (7.5) | 33.6 (6.4)

4. Primary Outcome: Caregiver: Quality of Life Measured With European Quality of Life (Euro-QOL)
Description: European Quality of Life (Euro--QL) measures 5 domains: mobility, self--care, usualactivities, pain/discomfort, and depression and have three levels of functioning each (no problems, some problems, and unable to/extreme problems). The VAS is a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: This was a 6-month study. We are reporting the change from baseline to the 6-month end of study time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
Number analyzed (Participants) | 24 | 22
score on a scale | 81.6 (11.1) | 70.8 (19.9)

5. Primary Outcome: Caregiver: Self Efficacy
Description: The self-efficacy score was a 8--item likert scale with each item rated from 1--5 (unable to most able). A total score for the instrument is provided by summing the scores of each item and dividing by the number of items producing a score in the range of 1-5. Higher overall mean scores indicate greater self efficacy.
Time Frame: This was a 6-month study. We are reporting the change from baseline to the 6-month end of study time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
Number analyzed (Participants) | 8 | 12
score on a scale | 4.4 (0.5) | 4.0 (0.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition does not differ from the clinicaltrials.gov definition. Participant enrollment includes caregivers and persons with dementia (PWD). While we had volunteers, they assisted with intervention delivery hence we did not collect any adverse events from them.
  Additionally, we have added a description to specify whether the AE was from a PWD or a caregiver.
Arm/Group | Treatment - Partners at Meals (PAM) | Enhanced Usual Condition (EUC)
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/21
Serious Adverse Events (participants affected / at risk) | 6/27 | 5/21
Other Adverse Events (participants affected / at risk) | 3/27 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment - Partners at Meals (PAM) (N=27) | Enhanced Usual Condition (EUC) (N=21)
Rectal bleeding - caregiver (Gastrointestinal disorders) | 1 (1) | 0 (0) — Only 1 caregiver reported this AE
Seizure - PWD (Nervous system disorders) | 1 (1) | 0 (0) — Only 1 PWD reported this AE
Dehydration - caregiver (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Only 1 caregiver reported this AE
Fall - PWD (Social circumstances) | 1 (1) | 0 (0) — Only 1 PWD reported this AE
Pneumonia - PWD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Only 1 PWD reported this AE
COVID - PWD (Infections and infestations) | 1 (1) | 1 (1) — Only 1 PWD reported this AE
Anemia - PWD (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Only 1 PWD reported this AE
Rash - PWD (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Only 1 PWD reported this AE
Arrhythmia and Heart Failure - PWD (Cardiac disorders) | 1 (1) | 1 (1) — Only 1 PWD reported this AE
Fainting - PWD (Nervous system disorders) | 1 (1) | 0 (0) — Only 1 PWD reported this AE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment - Partners at Meals (PAM) (N=27) | Enhanced Usual Condition (EUC) (N=21)
Muscle spasm - caregiver (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Only 1 caregiver reported this AE
COVID - PWD (Infections and infestations) | 3 (3) | 0 (0) — Only 3 PWDs reported this AE

LIMITATIONS AND CAVEATS:
Respite centers (from where the participants were recruited) shut down during the pandemic.

Sometimes participants wifi / internet access was limited Some caregivers expressed perceived burden of study procedures (e.g., taking pictures during mealtime and uploading) High staff / volunteer turnover in respite centers Lack of caregiver interest in participating in research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03622814/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03622814/ICF_001.pdf